CLINICAL TRIAL: NCT02025855
Title: Adjunct Methadone to Decrease the Duration of Mechanical Ventilation in the Medical Intensive Care Unit
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI no longer practicing at study institution.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Smoot_8503
Record Dates: First submitted 2013-12-30; First posted 2014-01-01 (Estimated); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use, Unspecified With Withdrawal; Opioid-Induced Disorders; Delirium
Keywords: Iatrogenic opioid abstinence syndrome; Methadone; Mechanical ventilation; ICU delirium; Continuous sedation
MeSH Terms: conditions — Delirium | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone (Experimental): Methadone will be administered at a dose calculated from the subjects total daily opioid requirements, with a maximum methadone dose of 60 mg per day. The methadone will be administered every 8 hours as 5 mg capsules that will be given via an enteral feeding tube.
  Interventions: Drug: Methadone
- Placebo (Placebo Comparator): This will be a capsule containing only lactose and will be given every 8 hours via an enteral feeding tube. The number of placebo capsules will be calculated based on the subjects opioid requirements. This will ensure the same number of capsules will be given despite which arm the patient is enrolled in.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methadone
  Arms: Methadone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if administering methadone to mechanically ventilated patients in the medical intensive care unit (ICU) requiring continuous infusions of sedatives and analgesics will decrease the time of mechanical ventilation, when initiated within 48 hours of their admission. Patients meeting enrollment criteria will be randomly assigned to receive methadone or placebo in addition to standard care. Methadone is a long acting pain medication that is approved by the Food and Drug Administration (FDA) to manage withdrawal from opioids and moderate to severe pain. Both of these indications are a frequent concern for critically ill patients that require mechanical ventilation. These patients often require intravenous (IV) opioids to manage the pain they experience due to their illness, procedures, and mechanical ventilation. During this time patients can develop physical dependence, which leads to withdrawal symptoms when the opioids are stopped or the dose is reduced. These symptoms can include agitation, pain, diarrhea and several others. Currently this is managed by a slow reduction in the dose of the IV opioid, but this can lead to prolonged time on mechanical ventilation, which has been associated with increased morbidity. Administering oral methadone to patients experiencing withdrawal symptoms has been shown to reduce and even eliminate these symptoms in the outpatient setting. This should also benefit patients in the ICU experiencing withdrawal from intravenous opioids required during their stay. It may allow for the other opioids to be discontinued more quickly, allowing for a shorter duration of mechanical ventilation.

The level of pain and sedation will be assessed between groups randomized to either methadone or placebo in addition to current intravenous sedative and analgesic agents. The duration of mechanical ventilation will be assessed between both groups. Opioid withdrawal symptoms may manifest or be mistaken for delirium symptoms. ICU delirium is often managed with antipsychotic medications. To assess if methadone can reduce the need for antipsychotic medication, all administered antipsychotic doses will be recorded and total consumption will be compared between the two groups. Methadone has been associated with abnormal heart rhythms in rare instances. To ensure patient safety, data from the heart monitor will be collected and compared between the two groups to assess for QT interval prolongation.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients with opioid consumption greater than or equal to 1,200 mcg of fentanyl or equivalent consumption of another opioid per day during the first 48 hours of intubation.

Exclusion Criteria:

* Allergy to methadone
* Admitted for head injury
* Admitted for seizure
* Seizure during admission, prior to enrollment
* Subjects at high risk for developing a prolonged corrected QT (QTc) interval
* Gastric residual volume ≥200 mL
* Suspected obstruction or ileus
* Nausea and vomiting
* Recent abdominal surgery
* Active upper or lower gastrointestinal bleeding
* Active order for no medications by mouth or Total parenteral nutrition (TPN)
* Pregnancy
* Subjects receiving neuromuscular blocker infusions
* Subjects taking antipsychotics at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Smoot, PharmD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Background] Kollef MH, Levy NT, Ahrens TS, Schaiff R, Prentice D, Sherman G. The use of continuous i.v. sedation is associated with prolongation of mechanical ventilation. Chest. 1998 Aug;114(2):541-8. doi: 10.1378/chest.114.2.541. PMID 9726743
- [Background] Wanzuita R, Poli-de-Figueiredo LF, Pfuetzenreiter F, Cavalcanti AB, Westphal GA. Replacement of fentanyl infusion by enteral methadone decreases the weaning time from mechanical ventilation: a randomized controlled trial. Crit Care. 2012 Dec 12;16(2):R49. doi: 10.1186/cc11250. PMID 22420584
- [Background] Lugo RA, MacLaren R, Cash J, Pribble CG, Vernon DD. Enteral methadone to expedite fentanyl discontinuation and prevent opioid abstinence syndrome in the PICU. Pharmacotherapy. 2001 Dec;21(12):1566-73. doi: 10.1592/phco.21.20.1566.34471. PMID 11765307
- [Background] Martell BA, Arnsten JH, Krantz MJ, Gourevitch MN. Impact of methadone treatment on cardiac repolarization and conduction in opioid users. Am J Cardiol. 2005 Apr 1;95(7):915-8. doi: 10.1016/j.amjcard.2004.11.055. PMID 15781034
- [Background] Tobias JD, Schleien CL, Haun SE. Methadone as treatment for iatrogenic narcotic dependency in pediatric intensive care unit patients. Crit Care Med. 1990 Nov;18(11):1292-3. doi: 10.1097/00003246-199011000-00024. No abstract available. PMID 1977561
- [Background] Johnson PN, Boyles KA, Miller JL. Selection of the initial methadone regimen for the management of iatrogenic opioid abstinence syndrome in critically ill children. Pharmacotherapy. 2012 Feb;32(2):148-57. doi: 10.1002/PHAR.1001. Epub 2012 Jan 24. PMID 22392424
- [Background] Bowens CD, Thompson JA, Thompson MT, Breitzka RL, Thompson DG, Sheeran PW. A trial of methadone tapering schedules in pediatric intensive care unit patients exposed to prolonged sedative infusions. Pediatr Crit Care Med. 2011 Sep;12(5):504-11. doi: 10.1097/PCC.0b013e3181fe38f5. PMID 21076361
- [Background] Hovav E, Weinstock M. Temporal factors influencing the development of acute tolerance to opiates. J Pharmacol Exp Ther. 1987 Jul;242(1):251-6. PMID 3612531

RESULTS

PARTICIPANT FLOW:
Groups:
- Methadone: Methadone will be administered at a dose calculated from the subjects total daily opioid requirements, with a maximum methadone dose of 60 mg per day. The methadone will be administered every 8 hours as 5 mg capsules that will be given via an enteral feeding tube.
  Methadone
- Placebo: This will be a capsule containing only lactose and will be given every 8 hours via an enteral feeding tube. The number of placebo capsules will be calculated based on the subjects opioid requirements. This will ensure the same number of capsules will be given despite which arm the patient is enrolled in.
  Placebo
Period: Overall Study
Arm/Group | Methadone | Placebo
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone | Placebo | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (14.9) | 37 (17.2) | 47 (19.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Time to Extubation
Description: The time to extubation will be calculated and compared for both groups.
Time Frame: Up to 14 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Methadone | Placebo
Number analyzed (Participants) | 4 | 5
Days | 10 [6.75 to 14] | 4 [4 to 6]

2. Secondary Outcome: Cumulative Opioid Consumption
Description: Cumulative doses of opioids will be collected and converted to morphine equivalents for analysis.
Time Frame: Up to 14 days
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalents
Arm/Group | Methadone | Placebo
Number analyzed (Participants) | 4 | 5
mg morphine equivalents | 473.5 [400 to 943] | 561 [514 to 2372]

3. Secondary Outcome: Level of Sedation
Description: Levels of pain and sedation will be assessed per institutional policy, which utilizes the Motor Agitation Assessment Scale (MAAS). Average daily scores will be collected and compared for each group. The MAAS is scored from 0 (patient unresponsive) to 6 (dangerously agitated, uncooperative patient).
Time Frame: Up to 14 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methadone | Placebo
Number analyzed (Participants) | 4 | 5
score on a scale | 3 [3 to 3] | 3 [3 to 3]

4. Secondary Outcome: Corrected QT Interval
Description: QTc intervals will be calculated and documented at baseline and every 24 hours after to ensure it does not become prolonged. These values will be compared between groups by taking the median of the baseline and daily values.
Time Frame: Up to 14 days
Measure: Median (Inter-Quartile Range); unit: ms
Arm/Group | Methadone | Placebo
Number analyzed (Participants) | 4 | 5
ms | 437 [430 to 439] | 457 [450 to 465]

5. Secondary Outcome: Cumulative Antipsychotic Use
Description: The number of doses of antipsychotic medications will be collected and compared as a surrogate marker for presumed delirium.
Time Frame: Up to 14 days
Measure: Median (Inter-Quartile Range); unit: doses
Arm/Group | Methadone | Placebo
Number analyzed (Participants) | 4 | 5
doses | 0 [0 to 2.25] | 0 [0 to 0]

6. Secondary Outcome: Cumulative Benzodiazepine Consumption
Description: Doses of all benzodiazepines will be collected and compared between groups to determine if methadone reduces consumption.
Time Frame: Up to 14 days
Measure: Median (Inter-Quartile Range); unit: mg midazolam
Arm/Group | Methadone | Placebo
Number analyzed (Participants) | 4 | 5
mg midazolam | 260 [119 to 408] | 445 [252.9 to 580]

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Methadone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol: Methadone Protocol (2014-11-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT02025855/Prot_000.pdf
  • Informed Consent Form: Methadone Informed Consent Form (2014-11-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT02025855/ICF_001.pdf